CLINICAL TRIAL: NCT05157360
Title: Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Sepsis Associated With Acute Necrotizing Soft Tissue Infections, The NASTI HAT Trial
Brief Title: HAT for the Treatment of Sepsis Associated With NASTI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow recruitment and not anticipated to meet recruitment numbers
Sponsor: Ascension Via Christi Hospitals Wichita, Inc. (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUVC1814
Record Dates: First submitted 2021-10-28; First posted 2021-12-15 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Necrotizing Soft Tissue Infection; Sepsis
MeSH Terms: conditions — Sepsis | interventions — Hydrocortisone; Ascorbic Acid; Thiamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: A randomization list will be used to show whether patients will be in group A or B. Only the Research Scientist who made the randomization list and the Pharmacy will know what group patients are in. The Burn Program Coordinator will get consent and enroll patients to the study. After that, the Burn Program Coordinator will call the pharmacy and report what group the patient is enrolled in, A or B. Then, the pharmacy will order the respective medications.
  The doctors and nurses providing care for the patients will not know who is in what treatment group, and neither will the patients.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm (Experimental): Patients will be enrolled within 24 hours of diagnosis of sepsis related to a necrotizing soft-tissue infections (NSTI). HAT will be initiated within 4 hours of enrollment (thus treatment with HAT can occur no later than 28 hours from diagnosis).
  Per Dr. Marik's original study, HAT consists of:
  1. 1.5 g vitamin C every 6 hours for 4 days or until ICU discharge
  2. 50 mg hydrocortisone every 6 hours for 7 days or until ICU discharge (followed by a taper over 3 days)
  3. 200 mg thiamine every 12 hours for 4 days or until ICU discharge In our study, due to the prolonged ICU course typical of most patients with NSTIs, it is not felt feasible to continue indefinitely "until ICU discharge." Thus, treatment will be continued for 4 to 7 days plus a 3 day taper (respectively) as above, with no plan for a longer duration of treatment.
  Interventions: Drug: HAT
- Control Arm (Placebo Comparator): The control arm will receive the same standard ICU care for NSTI but will not receive HAT. They will receive a placebo consisting of normal saline, indistinguishable to the treatment team (blinded) but known to the pharmacy team (unblinded to treatment and placebo groups). This is so that if the treatment team elects to give stress dose steroids, they can be administered without breaking protocol (i.e. if the patient is getting HAT, it includes steroids, so if the treating team wanted to start hydrocortisone - because they didn't know if the patient was on HAT or placebo and felt steroids were indicated - the pharmacist could ensure the patient was on steroids one way or another without unblinding the providers).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HAT — hydrocortisone, ascorbic acid (vitamin C), and thiamine (vitamin B1); referred to as HAT
  Other Names: hydrocortisone, vitamin C, vitamin B1
  Arms: Treatment Arm
Drug: Placebo — normal saline solution
  Other Names: NaCl 0.9%
  Arms: Control Arm

SUMMARY:
Evaluate the impact of HAT therapy versus placebo in the treatment of patients with an acute NSTI and sepsis.

DETAILED DESCRIPTION:
Primary outcome:

1. Hospital survival

Secondary outcomes:

1. Duration of vasopressor therapy
2. Requirement for renal replacement therapy in patients with Acute Kidney Injury (AKI)
3. ICU length of stay (LOS)
4. Change in serum procalcitonin (PCT) over first 72 hours
5. Change in SOFA score over first 72 hours (measured as SOFA score daily for four days, with day one being admission, then 3 days after, totaling 4 days of treatment with HAT)
6. Procalcitonin clearance (formula = initial PCT - 72 hour PCT divided by initial PCT x 100)
7. Number of wound related surgeries
8. Wound status at time of hospital discharge:

   1. Open
   2. Closed

ELIGIBILITY:
Inclusion Criteria:

1. Necrotizing soft tissue infection by clinical diagnosis and requiring surgical treatment.
2. Sepsis by clinical diagnosis and/or by Sepsis-3 criteria15, with source attributed to the wound.
3. Anticipated or confirmed intensive care unit

Exclusion Criteria: (Adapted from Sevransky et. al's VICTAS protocol)

1. Age < 18 years of age
2. Weight < 40 kg
3. Prior enrollment in this study or current enrollment in another study of any kind
4. Surgical findings, pathology/histology findings, or other findings determined to be inconsistent with an infectious acute NSTI such that the clinical diagnosis is no longer that of a NSTI
5. Sepsis deemed unlikely
6. Limitations of care during enrollment [defined as refusal of cardiovascular and respiratory support modes described in inclusion criteria, including "do not intubate" (DNI) status and comfort care]
7. Known allergy or known contraindication to vitamin C, thiamine, or corticosteroids [including previous history or active diagnosis of primary hyperoxaluria and/or oxalate nephropathy, or known/suspected ethylene glycol ingestion, or known glucose-6-phosphate dehydrogenase (G6PD) deficiency]
8. Use of vitamin C at a dose of >1g/day (IV or oral) within the 24 hours preceding first episode of qualifying organ dysfunction during a given Emergency Department or Intensive Care Unit admission
9. Chronic disease/illness that, in the opinion of the site investigator, have an expected lifespan of < 30 days unrelated to current sepsis diagnosis (e.g., stage IV malignancy, neurodegenerative disease, etc.)
10. Kidney Stone(s) of any kind
11. History of Oxalate Kidney Stone(s)
12. Pregnancy or known active breastfeeding
13. Prisoner or Incarceration
14. Inability or unwillingness of subject or legal surrogate/representative to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Resch, M.D., Principal Investigator — Surgeon
Locations (1):
- Ascension Via Christi Hospital - St. Francis Campus, Wichita, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Patients will be enrolled within 24 hours of diagnosis of sepsis related to a necrotizing soft-tissue infections (NSTI). HAT will be initiated within 4 hours of enrollment (thus treatment with HAT can occur no later than 28 hours from diagnosis).
  Per Dr. Marik's original study, HAT consists of:
  1. 1.5 g vitamin C every 6 hours for 4 days or until ICU discharge
  2. 50 mg hydrocortisone every 6 hours for 7 days or until ICU discharge (followed by a taper over 3 days)
  3. 200 mg thiamine every 12 hours for 4 days or until ICU discharge In our study, due to the prolonged ICU course typical of most patients with NSTIs, it is not felt feasible to continue indefinitely "until ICU discharge." Thus, treatment will be continued for 4 to 7 days plus a 3 day taper (respectively) as above, with no plan for a longer duration of treatment.
  HAT: hydrocortisone, ascorbic acid (vitamin C), and thiamine (vitamin B1); referred to as HAT
Period: Overall Study
Arm/Group | Treatment Arm | Control Arm
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.0 [50.5 to 68.0] | 54.0 [46.0 to 73.0] | 60.5 [46.8 to 67.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 4 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Hospital Survival
Description: Hospital survival is a binary variable showing whether the patient survived their time in the hospital. Hospital survival will be assessed from date of randomization until the date of discharge or date of death from any cause, whichever comes first, assessed up to 24 months.
Time Frame: Outcome is measured from date of admission to date of discharge or date of death, whichever comes first, approximately 7 to 10 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 5 | 5
Participants | 2 | 5

2. Secondary Outcome: Duration of Vasopressor Therapy
Description: The duration of vasopressor therapy is measured after date of randomization in hours and minutes from the initiation of vasopressor therapy until the termination of vasopressor therapy.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 5 | 5
hours | 53.8 [13.3 to 198.7] | 34.6 [14.7 to 88.0]

3. Secondary Outcome: Requirement for Renal Replacement Therapy in Patients With Acute Kidney Injury (AKI)
Description: This is a binary variable the will record whether the patient did or did not have a requirement for renal replacement therapy in patients with Acute Kidney Injury (AKI).
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

4. Secondary Outcome: ICU Length of Stay (LOS)
Description: ICU LOS will be measured by the date and time the patient was admitted to the ICU and by the date and time the patient was discharged from the ICU.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 5 | 5
days | 10.0 [7.5 to 12.0] | 7.0 [4.0 to 10.0]

5. Secondary Outcome: Change in Serum Procalcitonin (PCT) Over First 72 Hours
Description: This is a binary variable that will show whether there was a decrease in serum procalcitonin (PCT) over first 72 hours.
Time Frame: Over the first 72 hours from admission.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 5 | 5
Participants | 3 | 4

6. Secondary Outcome: Change in Sequential Organ Failure Assessment (SOFA) Score Over First 72 Hours (Measured as SOFA Score Daily for Four Days, With Day One Being Admission, Then 3 Days After, Totaling 4 Days of Treatment With HAT)
Description: This is a binary variable that will shows whether there was a decrease in SOFA score over the first 72 hours (measured as SOFA score daily for four days, with day one being admission, then 3 days after, totaling 4 days of treatment with HAT).
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 5 | 5
Participants | 4 | 5

7. Secondary Outcome: Procalcitonin Clearance
Description: Procalcitonin clearance (formula = initial PCT - 72 hour PCT divided by initial PCT x 100). The reported measure is median and range for those patients that
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: percentage of decrease in procalcitonin
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 5 | 5
percentage of decrease in procalcitonin | 23.5 [-23.6 to 78.2] | 77.9 [-655.6 to 83.8]

8. Secondary Outcome: Number of Wound Related Surgeries
Description: This is a variable that will show the count of wound related surgeries during the time the patient is admitted to the hospital.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Wound related surgeries
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 5 | 5
Wound related surgeries | 4.0 [2.5 to 4.0] | 2.0 [1.5 to 2.5]

9. Secondary Outcome: Wound Status at Time of Hospital Discharge: Open
Description: This shows the number of participants with an open wound at time of hospital discharge.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 5 | 5
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: From time of randomization until hospital discharge or death, whichever comes first. This time frame ranged from 7 to 10 days.
Arm/Group | Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 3/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Due to the small number of participants enrolled, the findings are observational only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT05157360/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT05157360/ICF_000.pdf